CLINICAL TRIAL: NCT01667159
Title: Adolescents With Major Depression and AUD: Community-Based Integrated Treatment
Brief Title: Community-Based Integrated Treatment for Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AA020705-01A1 (NIH); 1R01AA020705-01A1 (NIH)
Record Dates: First submitted 2012-08-14; First posted 2012-08-17 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Depression; Alcohol Use
Keywords: Depression; Alcohol Use; Outpatient Therapy
MeSH Terms: conditions — Depression; Alcohol Drinking | interventions — Standard of Care; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrated Cognitive Behavioral Therapy (Experimental): Adolescents and their parent(s) will receive integrated cognitive behavioral therapy.
  Interventions: Behavioral: Integrated Cognitive Behavioral Therapy
- Standard Care (Active Comparator): Adolescents and their parent(s) will receive treatment as usual through a community intensive outpatient program.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Integrated Cognitive Behavioral Therapy — Individual CBT sessions for parents and adolescents plus combined parent-adolescent family sessions delivered at least 1-2x each week for 6 months.
  Other Names: CBT for adolescents and parents
  Arms: Integrated Cognitive Behavioral Therapy
Behavioral: Standard Care — Intensive outpatient therapy with teens and their parents using a variety of eclectic treatments that characterize standard care for adolescents.
  Other Names: Intensive Outpatient Therapy; Treatment As Usual (TAU)
  Arms: Standard Care

SUMMARY:
This study will examine the effectiveness of an integrated treatment for adolescents who are depressed and use alcohol in an intensive outpatient setting in the community.

DETAILED DESCRIPTION:
Studies have consistently shown that alcohol use disorders (AUDs) and mental health disorders are related in adolescence. For example, in a community sample, teens who reported a history of AUD were almost four times as likely to have a history of Major Depressive Disorder (MDD) than teens with no history of AUD. The scientific community has only recently begun to examine how to treat adolescents with both AUD and MDD. Reviews have concluded that depression negatively affects treatment for substance abuse. At the same time, substance use issues are often not assessed or addressed in outpatient psychotherapy. Thus, we believe that protocols are needed to specifically address substance abusing, depressed adolescents. This study is designed to determine if an integrated (CBT-I) protocol designed to treat both substance use and depression in adolescents aged 12 to 18 years with AUD/MDD will produce better treatment outcomes compared to standard care (CBT-SC). Both the integrated CBT-I and CBT-SC conditions will be delivered by licensed mental health workers at a community mental health clinic - Gateway - that uses an Intensive Outpatient Program (IOP) model to treat adolescents with AUD and mental health disorders. Two hundred adolescents (50 per year for 4 years) will be recruited from Gateway's Dual Diagnosis IOP. If an adolescent screens in by reporting both depressed mood and substance abuse, these eligible families will complete a thorough baseline assessment and will then be assigned to either CBT-I or CBT-SC. The baseline battery will be repeated at the end of treatment, and 6 and 12 months after treatment completion to determine how families in the study do over time.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adolescent and parent
* Current substance use disorder
* Co-occurring psychiatric symptomatology

Exclusion Criteria:

* IQ < 80
* Diagnosis of psychotic disorder, pervasive developmental disorder, obsessive-compulsive disorder, bulimia nervosa or anorexia nervosa
* Adolescent use of illicit "hard" substances such as cocaine, heroine, and opiates 13 or more times over the prior 90 days

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Depression | Measured at 18 months from baseline

SECONDARY OUTCOMES:
Alcohol/Substance Use | Measured at 18 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Spirito A, Nestor B, Massing-Schaffer M, Esposito-Smythers C, Stout R, Frazier E, Gomez J, Graves H, Yen S, Hunt J, Wolff J. Predictors and moderators of marijuana and heavy alcohol use outcomes in adolescents treated for co-occurring substance use and psychiatric disorders in a randomized controlled trial. J Subst Abuse Treat. 2021 Dec;131:108536. doi: 10.1016/j.jsat.2021.108536. Epub 2021 Jun 15. PMID 34238628
- [Derived] MacPherson HA, Wolff J, Nestor B, Frazier E, Massing-Schaffer M, Graves H, Esposito-Smythers C, Spirito A. Parental Monitoring Predicts Depressive Symptom and Suicidal Ideation Outcomes in Adolescents Being Treated for Co-Occurring Substance Use and Psychiatric Disorders. J Affect Disord. 2021 Apr 1;284:190-198. doi: 10.1016/j.jad.2021.02.021. Epub 2021 Feb 9. PMID 33607509